CLINICAL TRIAL: NCT01035541
Title: Can Goal Directed Hemodynamic Management Improve Renal Outcome After Major Non-cardiac Surgery?
Brief Title: Goal Directed Hemodynamic Management and Renal Outcome After Major Non-cardiac Surgery
Acronym: IROM
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: IROM
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Major Non-cardiac Surgery
Keywords: Major non-cardiac surgery,; hemodynamic management,; PiCCO,; acute kidney injury,; renal outcome
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- P group: Fluid Management according to measurements with PiCCO®
  Interventions: Device: PiCCO® Monitoring
- C group: Conventional fluid management
  Interventions: Device: PiCCO® Monitoring

INTERVENTIONS:
Device: PiCCO® Monitoring — Fluid and vasopressor management according to PiCCO measruements

SUMMARY:
This study is designed to compare renal outcome of patients following major non-cardiac surgery with different perioperative hemodynamic managements: a goal directed hemodynamic management group (using PiCCO) and a control group.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication after major surgery. Many studies showed that AKI is associated with different complications: higher mortality, renal replacement therapy and prolonged hospital stay resulting in higher health care costs.

Until now just a few studies are published on prevention or therapy of AKI after major surgery. Most of these investigations are underpowered or show just marginal benefit. There are no studies published investigating the impact of goal-directed hemodynamic management on renal outcome following non-cardiac major surgery, even though hemodynamic stability seems to be of paramount importance for the kidneys.

Aim of this study is to investigate the impact of a goal directed hemodynamic management on renal outcome after major non-cardiac surgery.

Therefore patients will be randomized in one of two groups, the PiCCO group with goal directed hemodynamic management and the Control group, where PICCO data will be collected but will not influence hemodynamic management. In both groups the monitoring with transpulmonary thermodilution will be continued in the intensive care unit until 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective major non-cardiac surgery lasting more than 3 hours with a following intensive care unit stay for more than 3 days:

  * gastrectomy
  * pancreas surgery
  * small bowel surgery
  * esophageal surgery
* Age ≥ 18 years
* ASA classification I to III
* Written informed consent

Exclusion Criteria:

* Need for dialysis
* Contraindications for an arterial line in the femoral artery:

  * stents
  * bypasses
  * severe peripheral artery occlusive disease
* ASA classification IV to V
* Pregnant Woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients udndergoing Major non-cardiac surgery
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
maximum change in serum creatinine within 3 days | Start of anesthesia until third postoperative day (72 hours)

SECONDARY OUTCOMES:
incidence of AKI according to the RIFLE criteria, need for dialysis, pulmonal complications, rate of anastomotic insufficiency, sepsis, reoperation | 1 year
  All points are additionnally registered one year after the operation via telephone-questionnaire of the patient and his general practitioner

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Goepfert MS, Reuter DA, Akyol D, Lamm P, Kilger E, Goetz AE. Goal-directed fluid management reduces vasopressor and catecholamine use in cardiac surgery patients. Intensive Care Med. 2007 Jan;33(1):96-103. doi: 10.1007/s00134-006-0404-2. Epub 2006 Nov 21. PMID 17119923
- [Derived] Schmid S, Kapfer B, Heim M, Bogdanski R, Anetsberger A, Blobner M, Jungwirth B. Algorithm-guided goal-directed haemodynamic therapy does not improve renal function after major abdominal surgery compared to good standard clinical care: a prospective randomised trial. Crit Care. 2016 Mar 8;20:50. doi: 10.1186/s13054-016-1237-1. PMID 26951105